CLINICAL TRIAL: NCT03675815
Title: Body Composition Sub-study of the D2EFT Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2EFT BodyComp
Record Dates: First submitted 2018-07-02; First posted 2018-09-18 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Tablets; Ritonavir; Nucleosides; dolutegravir; Tenofovir; Lamivudine; Racivir; Capsules; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of care (Active Comparator): darunavir 800 mg oral tablet + ritonavir 100 mg oral tablet + (N(t)RTIs) po qd
  Interventions: Drug: Darunavir (DRV) 800 milligram (MG) Oral Tablet; Drug: Ritonavir 100 MG Oral Tablet; Drug: N(t)RTIs
- Dolutegravir + tenofovir (TDF) + either lamivudine (3TC) or emtricitabine (FTC) (Experimental): dolutegravir 50 mg oral tablet + TDF 300 mg oral tablet + either 3TC 300 mg oral tablet or FTC 200 mg oral capsule po qd
  Interventions: Drug: Dolutegravir 50 MG Oral Tablet; Drug: TDF 300 MG Oral Tablet; Drug: 3TC 300 MG Oral Tablet; Drug: FTC 200 MG Oral Cap
- Dolutegravir + darunavir (Experimental): dolutegravir 50 mg oral tablet + darunavir 800 mg oral tablet + ritonavir 100 mg oral tablet po qd
  Interventions: Drug: Darunavir (DRV) 800 milligram (MG) Oral Tablet; Drug: Ritonavir 100 MG Oral Tablet; Drug: Dolutegravir 50 MG Oral Tablet

INTERVENTIONS:
Drug: Darunavir (DRV) 800 milligram (MG) Oral Tablet — 800 milligrams (mg) orally once daily for 96 weeks
  Other Names: Prezista
  Arms: Dolutegravir + darunavir; Standard of care
Drug: Ritonavir 100 MG Oral Tablet — 100 mg orally once daily for 96 weeks
  Other Names: Norvir, RTV
  Arms: Dolutegravir + darunavir; Standard of care
Drug: N(t)RTIs — Choice of N(t)RTIs determined by clinician guided by either genotypic resistance testing or use of a protocol-specified algorithm for N(t)RTI selection
  Other Names: Nucleoside/nucleotide reverse transcriptase inhibitors [N(t)RTIs]
  Arms: Standard of care
Drug: Dolutegravir 50 MG Oral Tablet — 50 mg orally once daily for 96 weeks
  Other Names: Tivicay, DTG
  Arms: Dolutegravir + darunavir; Dolutegravir + tenofovir (TDF) + either lamivudine (3TC) or emtricitabine (FTC)
Drug: TDF 300 MG Oral Tablet — 300 mg orally once daily for 96 weeks
  Other Names: tenofovir disoproxil fumarate, Viread
  Arms: Dolutegravir + tenofovir (TDF) + either lamivudine (3TC) or emtricitabine (FTC)
Drug: 3TC 300 MG Oral Tablet — 300 mg orally once daily for 96 weeks. Choice of 3TC or FTC will be determined by clinician
  Other Names: lamivudine
  Arms: Dolutegravir + tenofovir (TDF) + either lamivudine (3TC) or emtricitabine (FTC)
Drug: FTC 200 MG Oral Cap — 200 mg orally once daily for 96 weeks. Choice of emtricitabine or lamivudine will be determined by clinician
  Other Names: Emtriva, emtricitabine
  Arms: Dolutegravir + tenofovir (TDF) + either lamivudine (3TC) or emtricitabine (FTC)

SUMMARY:
This is a non-randomised, controlled, parallel group, sub-study of D2EFT (NCT03017872), a randomised, open-label study in approximately 1,000 HIV-infected adults failing first-line antiretroviral therapy (ART) in low-middle income countries. The sub-study will be offered to all D2EFT sites with access to DXA technology for whole-body composition analysis. Sites will offer the sub-study to consecutive clinic patients. Patients must be approached for participation and provide informed written consent prior to randomisation into D2EFT. This study will recruit approximately 300 patients. Allocation to one of three ART treatment regimens will follow the result of D2EFT randomisation. The study will investigate the role of contemporary ART on body composition and metabolic parameters by comparing over 96 weeks the effects of the D2EFT ART regimens. The primary endpoint will be assessed at week 48.

DETAILED DESCRIPTION:
Consenting participants will be randomised within the main D2EFT protocol to receive either ritonavir-boosted darunavir plus two nucleosides or dolutegravir plus two predetermined nucleosides (lamivudine or emtricitabine) or ritonavir-boosted darunavir plus dolutegravir. Enrolment into the sub-study is voluntary and not a requirement for enrolment into D2EFT. Parameters relevant to this study including demographics, arm of randomised ART, smoking status, body habitus and fasting lipid parameters and resting blood pressure at required time points will be collected as part of the main D2EFT study. Sub-study specific assessments performed at baseline and at weeks 48 and 96 include clinical and laboratory assessments, sample collection and dual-energy X-ray absorptiometry (DXA)-assessed whole-body composition. Consenting participants will have blood for storage collected at weeks 0, 48 and 96. The specimens will be used for future studies into treatment of HIV infection and immunity.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil the criteria for D2EFT randomisation
* Able to undergo DXA whole-body scanning
* Provide informed written consent for the D2EFT Body Composition Sub-study

Exclusion Criteria:

* Unwilling to comply with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Mean/median between-group change in waist-to-hip ratio | at 48 weeks
  umbilical waist and hip measures
Mean/median between-group change in total-to-HDL cholesterol ratio | at 48 weeks
  total and HDL cholesterol plasma concentrations

SECONDARY OUTCOMES:
Mean/median between-group change in total-to-HDL cholesterol ratio | at 96 weeks
  total and HDL cholesterol plasma concentrations
Mean/median between-group change in waist-to-hip ratio | at 96 weeks
  umbilical waist and hip measures
Mean/median between-group change in body weight | at week 48 and 96
  body weight measurement
Mean/median between-group change in maximum umbilical and hip measures | at week 48 and 96
  umbilical waist and hip measures
Mean/median between-group change in fasting lipid parameters | at weeks 48 and 96
  total, HDL, and LDL cholesterol and triglyceride plasma concentrations
Mean/median between-group change in fasting glycaemic parameters | at weeks 48 and 96
  glucose, insulin, HbA1c concentrations
Mean/median between-group absolute change in limb fat assessed by DXA | week 48 and 96
  absolute change from baseline in limb fat
Mean/median between-group percentage change in limb fat assessed by DXA | week 48 and 96
  percentage change from baseline in limb fat
Mean/median between-group changes in regional body fat assessed by DXA | week 48 and 96
  regional = limb fat and truncal fat
Mean/median between-group changes in total body fat and lean tissue assessed by DXA | week 48 and 96
  total body fat and total lean tissue
Mean/median between-group changes in bone mineral content assessed by DXA | week 48 and 96
  total bone mineral content
Mean/median between-group change in Body Image questionnaire scores | weeks 48 and 96
  NIAID Adult AIDS Clinical Trials Group Baseline and Follow-up questionnaires
Proportion with Metabolic Syndrome | week 0, and week 48 and 96
  baseline prevalence and incidence at weeks 48 and 96

OTHER OUTCOMES:
Mean/median between-group change in serum biomarker concentrations | weeks 48 and 96
  biomarkers to be determined

CONTACTS AND LOCATIONS:
Overall Officials: Gail Matthews, MBBCh, Principal Investigator — The Kirby Institute, UNSW Sydney
Locations (7):
- Chennai Antiviral Research aznd Treatment (CART) Clinical Research Site, Chennai, India
- Univerity of Malaya Medical Centre, Kuala Lumpur, Malaysia
- South Africa (3):
  - Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital, Soweto, Johannesburg
  - Clinical HIV Research Unit, Helen Joseph Hospital, Westdene, Johannesburg
  - Desmond Tutu HIV Foundation, Cape Town
- The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Thai Red Cross Research Centre, Bangkok, Thailand
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe